CLINICAL TRIAL: NCT02954978
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of Low Doses of Nilotinib Treatment on Safety, Tolerability, Pharmacokinetics and Biomarkers in Parkinson's Disease
Brief Title: Impact of Nilotinib on Safety, Tolerability, Pharmacokinetics and Biomarkers in Parkinson's Disease
Acronym: PD Nilotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Fernando Pagan MD, Associate Professor, Department of Neurology Co-Director, Movement Disorders Program Director, NPF Center of Excellence Associate Professor, SOM Clinical Track, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB# 2016-0380
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease; Parkinsons Disease With Dementia
MeSH Terms: conditions — Parkinson Disease | interventions — nilotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Out of seventy five (75) participants that will be recruited and randomly assigned 1:1:1 to the three (3) groups (arms), 25 patients in group 1 will receive the placebo ("sugar pill") one (1) capsule by mouth once daily (taken without a meal) for 12 months and 3 months follow up.
  Interventions: Drug: Placebo Oral Capsule
- Nilotinib 150mg (Active Comparator): Out of seventy five (75) participants that will be recruited and randomly assigned 1:1:1 to the three (3) groups (arms), 25 patients in group 2 will receive 150mg Nilotinib one (1) capsule once daily (taken without a meal) for 12 months and 3 months follow up.
  Interventions: Drug: Nilotinib 150mg oral capsule [Tasigna]
- Nilotinib 300mg (Active Comparator): Out of seventy five (75) participants that will be recruited and randomly assigned 1:1:1 to the three (3) groups (arms), 25 patients in group 3 will receive 300mg Nilotinib one (1) capsule once daily (taken without a meal) for 12 months and 3 months follow up.
  Interventions: Drug: Nilotinib 300mg oral capsule [Tasigna]

INTERVENTIONS:
Drug: Placebo Oral Capsule — 25 patients in group 1 will receive Placebo ("sugar pill") one (1) capsule once daily (taken without a meal) for 12 months and 3 months follow up.
  Other Names: Placebo
  Arms: Placebo
Drug: Nilotinib 150mg oral capsule [Tasigna] — 25 patients in group 2 will receive 150mg Nilotinib one (1) capsule once daily (taken without a meal) for 12 months and 3 months follow up.
  Other Names: Nilotinib low dose
  Arms: Nilotinib 150mg
Drug: Nilotinib 300mg oral capsule [Tasigna] — 25 patients in group 3 will receive 300mg Nilotinib one (1) capsule once daily (taken without a meal) for 12 months and 3 months follow up.
  Other Names: Nilotinib high dose
  Arms: Nilotinib 300mg

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disorder causing motor and non-motor symptoms. PD is characterized by death of dopaminergic (DA) neurons in the substantia nigra (SN) pars compacta and formation of inclusions known as Lewy bodies (LBs) that primarily contain aggregated alpha-Synuclein. Nilotinib (Tasigna®, AMN107, Novartis, Switzerland) is approved by U.S. Food and Drug Administration (FDA) and is well tolerated for CML treatment at oral doses of 600-800mg daily. Nilotinib penetrates the brain and promotes autophagic degradation of alpha-Synuclein and p-Tau, leading to survival of DA neurons and improvement of motor function in PD models. For these studies, Nilotinib (1-10mg/kg daily) was used at significantly less than the clinically approved dose (up to 1200mg daily) in CML.

DETAILED DESCRIPTION:
Based on strong pre-clinical evidence of the effects of Nilotinib on neurodegenerative pathologies, including autophagic clearance of neurotoxic proteins, neurotransmitters (dopamine and glutamate), immunity and behavior, the investigators conducted an open label pilot clinical trial in advanced PD with dementia (PDD) and Dementia with Lewy Body (DLB) (stage 3-4) patients. Participants (N=12) were randomized 1:1 to once daily oral dose of 150mg and 300mg Nilotinib for 6 months. The investigators' data suggest that Nilotinib penetrates the brain and inhibits CSF Abelson (Abl) activity via reduction of phosphorylated Abl in agreement with pre-clinical data. Several studies show that CSF alpha-Synuclein and Abeta42 are decreased and CSF total Tau and p-Tau are increased in PD and DLB. The investigators' data show attenuation of loss of CSF alpha-Synuclein and Abeta40/42 with 300mg (50% of the CML dose) compared to 150mg Nilotinib after 6 months treatment. CSF homovanillic acid (HVA), which is an end by-product of dopamine, is significantly increased; and CSF total Tau and p-Tau are significantly reduced (N=5, P<0.05) with 300mg Nilotinib between baseline and 6 months treatment. Despite the reduction of L-Dopa replacement therapies in our study, UDPRS I-IV scores improved with 150mg (3.5 points) and 300mg (11 points) from baseline to 6 months and worsened (13.7 points and 11.4 points) after 3 months withdrawal of 150mg and 300mg, respectively. Other non-motor functions e.g. constipation was resolved in all patients and cognition was also improved (3.5 points) using both the Mini-Mental Status Exam (MMSE) or the Scales for Outcomes in Parkinson's Disease-Cognition (SCOPA-Cog) between baseline and 6 months. MMSE scores returned to baseline after 3 months of Nilotinib withdrawal. These data are very compelling to evaluate the effects of Nilotinib in a phase II, randomized, double-blind, placebo-controlled trial in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative (LAR).
3. Patients between the age of 40-90 years, medically stable
4. Diagnosis of PD according to the UK Brain Bank Diagnostic Criteria
5. PD subjects with MoCA ≥ 22
6. 2.5 ≥Hoehn and Yahr stage ≤3
7. No mono-amine oxidase (MAO)-B inhibitors (Selegeline or rasagiline) are allowed at least 6 weeks before enrollment
8. Must be medically stable on 800mg Levodopa daily for at least 4 weeks
9. QTc interval 350-460 ms, inclusive
10. Participants must be willing to undergo LP at baseline and 12 months after treatment

Exclusion Criteria:

1. Patients with hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥461 ms
2. Concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infraction or cardiac failure, angina, arrhythmia
3. History or presence of cardiac conditions including:

   * Cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke)
   * Congestive heart failure
   * First, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
   * Any history of Torsade de Pointes
4. Treatment with any of the following drugs at the time of screening or the preceding 30 days, and/or planned use over the course of the trial:

   * Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine)
   * Treatment with QT prolonging drugs (www.crediblemeds.org)- excluding Selective Serotonin Reuptake Inhibitors (SSRIs) (e.g. Citalopram, Paxil, Zoloft, Cymbalta, Sertraline, etc...)
   * Strong CYP3A4 inhibitors (including grapefruit juice). The concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole) must be avoided. Grapefruit products may also increase serum concentrations of Nilotinib. Should treatment with any of these agents be required, therapy with Nilotinib should be interrupted.
   * Anticoagulants, including Coumadin (warfarin), heparin, enoxaparin, daltiparin, xarelto, etc.
   * St. John's Wort and the concomitant use of strong other CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) must be avoided since these agents may reduce the concentration of Nilotinib.
5. Abnormal liver function defined as AST and/or ALT > 100% the upper limit of the normal
6. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
7. History of HIV, clinically significant chronic hepatitis, or other active infection
8. Females must not be lactating, pregnant or with possible pregnancy
9. Medical history of liver or pancreatic disease
10. Clinical signs indicating syndromes other than idiopathic PD, including corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, Babinski sign
11. Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
12. Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality
13. Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of skin melanoma or stable prostate cancer are not exclusionary)
14. Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder
15. Must not be on any immunosuppressant medications (e.g. IVig)
16. Must not be enrolled as an active participant in another clinical study
17. Diagnosis of DLB

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Safety will be measured by number of participants experiencing the occurrence of adverse events and/or abnormal laboratory values | 12 months
  Safety will be measured by assessing number of participants with abnormal laboratory values, as well as adverse events (AEs) and serious adverse events (SAEs) deemed to be possibly, probably, or definitely related to the study drug.

SECONDARY OUTCOMES:
Effects of nilotinib treatment on levels of homovanillic acid in cerebrospinal fluid | 12 months
  The investigators will determine the effects of nilotinib on cerebrospinal fluid levels of homovanillic acid between baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Pagan, MD, Principal Investigator — Georgetown University
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pagan F, Hebron M, Valadez EH, Torres-Yaghi Y, Huang X, Mills RR, Wilmarth BM, Howard H, Dunn C, Carlson A, Lawler A, Rogers SL, Falconer RA, Ahn J, Li Z, Moussa C. Nilotinib Effects in Parkinson's disease and Dementia with Lewy bodies. J Parkinsons Dis. 2016 Jul 11;6(3):503-17. doi: 10.3233/JPD-160867. PMID 27434297
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102
- [Derived] Fowler AJ, Ahn J, Hebron M, Chiu T, Ayoub R, Mulki S, Ressom H, Torres-Yaghi Y, Wilmarth B, Pagan FL, Moussa C. CSF MicroRNAs Reveal Impairment of Angiogenesis and Autophagy in Parkinson Disease. Neurol Genet. 2021 Nov 12;7(6):e633. doi: 10.1212/NXG.0000000000000633. eCollection 2021 Dec. PMID 34786477
- [Derived] Pagan FL, Hebron ML, Wilmarth B, Torres-Yaghi Y, Lawler A, Mundel EE, Yusuf N, Starr NJ, Anjum M, Arellano J, Howard HH, Shi W, Mulki S, Kurd-Misto T, Matar S, Liu X, Ahn J, Moussa C. Nilotinib Effects on Safety, Tolerability, and Potential Biomarkers in Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2020 Mar 1;77(3):309-317. doi: 10.1001/jamaneurol.2019.4200. PMID 31841599
- See also: https://sites.google.com/a/georgetown.edu/moussa-lab/home3 — https://neurology.georgetown.edu/translational_neurotherapeutics